CLINICAL TRIAL: NCT03190876
Title: Prevention of Seroma Formation After Body Contouring Procedures
Brief Title: Seroma Prevention After Body Contouring Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Dr. Alexandra Anker, Principal Investigator, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-101-0292
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Seroma; Abdominoplasty; Complication of Surgical Procedure
Keywords: Drain usage
MeSH Terms: conditions — Seroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Suction drain (No Intervention): Conventional body contouring procedure, application of Redon suction drains, drain removal when output is less than 30 ml in 24 hours or at the latest on postoperative day 7
- Passive drain (Active Comparator): Conventional body contouring procedure, application of drains without suction (passive drainage), drain removal when output is less than 30 ml in 24 hours or at the latest on postoperative day 7
  Interventions: Procedure: Variable drain usage
- No drain (Active Comparator): Conventional body contouring procedure, no application of drains
  Interventions: Procedure: Variable drain usage

INTERVENTIONS:
Procedure: Variable drain usage — Influence of drain usage on seroma formation rate
  Arms: No drain; Passive drain

SUMMARY:
With a prevalence of up to 25%, seroma formation is among the most common complications of body contouring procedures such as abdominoplasty. Small amounts of fluid are reabsorbed by the body spontaneously, however, larger seroma volumes need to be evacuated via puncture aspiration to prevent wound healing disturbances and infection, leading to major patient discomfort and a prolonged hospital stay. There is increasing controversy regarding the efficacy of surgical drains in seroma prevention. This study compares the incidence rate of seroma in three study arms with different usage of drains.

ELIGIBILITY:
Inclusion Criteria:

* All full-aged patients requiring body contouring procedures in our department who provide oral and written informed consent indicating that they agree to participate in the study

Exclusion Criteria:

* Minors or patients with a designated health care proxy, revision surgeries, morbid obesity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of seroma formation | Weekly follow-up until postoperative week 6.
  As primary outcome this study measures the rate of seroma requiring evacuation via puncture aspiration (fluid retention > 20 cc) in each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Plastic Surgery, University Hospital of Regensburg, Regensburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No